CLINICAL TRIAL: NCT04555330
Title: Technology Assisted Physical Activity Among Hospitalised Medical Patients
Acronym: TAPAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FYS-2019-017
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease; Cardiac Disease; Geriatric Disease
MeSH Terms: conditions — Lung Diseases; Heart Diseases

STUDY DESIGN:
Intervention Model Description: The allocation of participants will be done in 8 waves at each of the participating wards. At each hospital ward, 4 of the waves will be allocated to the control group and 4 to the intervention group. The order of the conditions is randomised.
  A participant will be assigned to the wave that the ward is allocated to at the time of admission.
  The wave size for each ward is set to 10 patients.
  Assignment of the waves at each department will be determined before any recruitment by means of Latin square randomisation in 2 blocks of 4 waves at the 4 participating wards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Feedback (Experimental): Participants in the intervention group will receive usual hospital care and be provided with a sensor collecting data on physical activity level during hospitalisation AND a monitor placed at their bedside that displays information about their physical activity level and motivation to move. This information will be visible to the health personnel, the patients and visitors.
  Interventions: Device: Physical activity measurement; Device: Visual Feedback
- Control Group (Other): The participants in the non-exposed cohort will receive usual hospital care and be provided with a sensor collecting data on activity level during hospitalisation.No feedback on physical activity is provided.
  Interventions: Device: Physical activity measurement

INTERVENTIONS:
Device: Physical activity measurement — To assess physical activity two small tri-axial accelerometers embedded in medical Band-Aids will be used. The accelerometers are discretely worn on the lateral aspect of the thigh.
  The accelerometers sample accelerations continuously during hospitalisation and are connected wirelessly to a tablet that via an inbuilt algorithm classify the recordings as bedridden (lying down), sitting, standing, and walking.
Device: Visual Feedback — The tablet will be placed on the patients bedside table and provides feedback on the amount of physical activity and motivational imagesand texts that will be visible for the patients, the health care staff and visitors.
  Arms: Visual Feedback

SUMMARY:
Research show that inactivity during hospitalization is the norm and that the negative effects on muscle mass and the fitness of the patient will take a long time and hard work to recover afterwards.

Especially for weaker elderly patients, just a few days in bed could mean that they are not able to take care of themselves afterwards, with increased care expenses and increased risk of relapse as a consequence. Even though this is known, the work to motivate patients to be active during their hospitalization is limited to few training sessions with only the most vulnerable patients. No tools are today available for objectively tracking and motivating patients to be active during their stay. Having such a professional tool would not only motivate but also shift the attention of the health professionals towards the importance of physical activity in the treatment of the patient.

The aim of the studys is to investigate if patients hospitalised for medical disease will increase their time spent out of bed during hospitalisation through simple visual feedback about physical activities from a mobile bedside device.

DETAILED DESCRIPTION:
The study will be conducted as a quasi-randomised trial using a large tertiary public hospital in Copenhagen, Denmark. Patients admitted to Department of Respiratory Medicine (2 wards), Department of Cardiology, and Department of Geriatrics will be included, and they will have their physical activity level measured either with or without a bedside monitor providing visual feedback of time spent bedridden, sitting, standing and walking.

All participants will have their physical activity measured during hospitalisation. Approximately half of the participants will receive visual feedback about the amount of physical activity from a mobile device placed on the bedside table.

ELIGIBILITY:
INCLUSION CRITERIA

An individual will be eligible for study participation if he/she meets the following criteria:

1. Is admitted to one of the participating departments
2. Has signed informed consent
3. Reads and speaks Danish

EXCLUSION CRITERIA

An individual will be excluded from the study if he/she meets any of the following criteria:

1. Any condition that, in the opinion of the investigator, makes the person unfit for participation
2. Expected hospitalisation less than 24 hours
3. Has no independent ambulatory abilities (e.g. wheel chair user)
4. Needs personal assistance in body transfers and ambulation (Cumulated Ambulation Score 0, 1, 2, or 3)
5. Has allergy towards band aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2016-06-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Time spent out of bed measured in minutes related to the total accelerometer wear time (minutes). | Through hospital stay, on average between 1 and 7 days

SECONDARY OUTCOMES:
Time spent lying down, measured in minutes related to the total accelerometer wear time (minutes). | Through hospital stay, on average between 1 and 7 days
Time spent sitting measured in minutes related to the total accelerometer wear time (minutes). | Through hospital stay, on average between 1 and 7 days
Time spent standing measured in minutes related to the total accelerometer wear time (minutes). | Through hospital stay, on average between 1 and 7 days
Time spent walking measured in minutes related to the total accelerometer wear time (minutes). | Through hospital stay, on average between 1 and 7 days
Length of stay | Time from hospital admission to hospital discharge
  Length of hospitalisation measured in days
Readmission to hospital | within 90 days
In-hospital fall incidents | Through hospital stay, on average between 1 and 7 days
  Number of falls recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request sen to the sponsor and/or invesitgators